CLINICAL TRIAL: NCT04838990
Title: TELE MS RCT: A Randomized Controlled Trial to Evaluate Feasibility of Remote Patient Visits in People With Multiple Sclerosis
Brief Title: TELEMS: Feasibility of Remote Patient Visits in MS
Acronym: TELEMSRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Patrick Altmann MD PhD, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2157/2020
Record Dates: First submitted 2021-02-21; First posted 2021-04-09 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; remote visits; telemedicine; remote patient monitoring; remote monitoring
MeSH Terms: conditions — Multiple Sclerosis | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional visit (Active Comparator): Regular outpatient visit
  Interventions: Other: EDSS; Other: Discussion of symptoms, Patient reported outcome (MSIS)
- phone visit (Experimental): Remote visit via phone
  Interventions: Other: EDSS; Other: Discussion of symptoms, Patient reported outcome (MSIS)
- video visit (Experimental): Remote visit via videochat
  Interventions: Other: EDSS; Other: Discussion of symptoms, Patient reported outcome (MSIS)

INTERVENTIONS:
Other: EDSS — Neurological Exam - EDSS (Expanded Disability Status Scale)
Other: Discussion of symptoms, Patient reported outcome (MSIS) — Patients will be asked about their wellbeing

SUMMARY:
This trials randomizes patients with multiple sclerosis (MS, pwMS) to a remote visit (via phone or videochat) or a regular outpatient visit. Outcomes include satisfaction on the patients' and doctor's side.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of any type of MS
* own a phone/smartphone/computer
* informed consent

Exclusion Criteria:

* language barriers

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
TMPQ | 1 week after intervention
  Telemedicine Perception questionnaire (17-85, higher scores are better)

SECONDARY OUTCOMES:
PPSM | 1 week after intervention
  Patient and Physician Satisfaction with monitoring (6-30, higher scores are better)

OTHER OUTCOMES:
Ancillary Analyses | immediately after the intervention
  Subgroup analyses comparing scores on the TMPQ above and below the median (Telemedicine Perception questionnaire, 17-85 points, higher scores are better) with clinical characteristics (EDSS and MSIS and Age)
Empirical Questionnaire | 1 week after intervention
  Participants are given an opportunity to openly provide feedback

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Altmann, MD PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request and through our local ERB.
Supporting Information: Study Protocol, ICF
Time Frame: Upon request and for 1 month
Access Criteria: reasonable request and upon approval of our local ERB

REFERENCES:
- [Derived] Altmann P, Leutmezer F, Ponleitner M, Ivkic D, Krajnc N, Rommer PS, Berger T, Bsteh G. Remote visits for people with multiple sclerosis during the COVID-19 pandemic in Austria: The TELE MS randomized controlled trial. Digit Health. 2022 Jul 11;8:20552076221112154. doi: 10.1177/20552076221112154. eCollection 2022 Jan-Dec. PMID 35847524